CLINICAL TRIAL: NCT03032380
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Clinical Study of S-649266 Compared With Meropenem for the Treatment of Hospital-acquired Bacterial Pneumonia, Ventilator-associated Bacterial Pneumonia, or Healthcare-associated Bacterial Pneumonia Caused by Gram-negative Pathogens
Brief Title: Clinical Study of Cefiderocol (S-649266) for the Treatment of Nosocomial Pneumonia Caused by Gram-negative Pathogens
Acronym: APEKS-NP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1615R2132; 2016-003020-23 (EudraCT Number)
Expanded Access: NCT03780140 (Approved for marketing)
Record Dates: First submitted 2017-01-17; First posted 2017-01-26 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Healthcare-associated Pneumonia (HCAP); Hospital Acquired Pneumonia (HAP); Ventilator Associated Pneumonia (VAP)
Keywords: Hospital-acquired pneumonia (HAP); S-649266; linezolid; meropenem; Healthcare-associated pneumonia (HCAP); nosocomial pneumonia; Ventilator-associated pneumonia (VAP); Gram-negative pathogens; pneumonia; cefiderocol
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated; Pneumonia | interventions — Cefiderocol; Meropenem; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cefiderocol (Experimental): Participants will receive 2 g cefiderocol administered intravenously every 8 hours for 7 to 14 days and 600 mg linezolid administered intravenously every 12 hours for at least 5 days.
  Interventions: Drug: Cefiderocol; Drug: Linezolid
- Meropenem (Active Comparator): Participants will receive 2 g meropenem administered intravenously every 8 hours for 7 to 14 days and 600 mg linezolid administered intravenously every 12 hours for at least 5 days.
  Interventions: Drug: Meropenem; Drug: Linezolid

INTERVENTIONS:
Drug: Cefiderocol — 2000 mg intravenously every 8 hours for a period of 7 to14 days (dosage adjustment is necessary based on renal function)
  Other Names: S-649266
  Arms: Cefiderocol
Drug: Meropenem — 2000 mg intravenously every 8 hours for a period of 7 to 14 days (dosage adjustment is necessary based on renal function)
  Other Names: Merrem®
  Arms: Meropenem
Drug: Linezolid — 600 mg of linezolid administered intravenously over 30 minutes to 2 hours, every 12 hours.
  Other Names: Zyvox®

SUMMARY:
The primary objective of this study is to compare all-cause mortality at Day 14 in participants receiving cefiderocol with participants receiving the comparator, meropenem, in adults with hospital-acquired bacterial pneumonia (HABP), ventilator-associated bacterial pneumonia (VABP), or healthcare-associated bacterial pneumonia (HCABP) caused by Gram-negative pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years or older at the time of signing informed consent
* Subjects who have provided written informed consent or their informed consent has been provided by a legally authorized representative
* Subjects who meet the clinical diagnosis criteria for hospital-acquired bacterial pneumonia (HABP), ventilator-associated bacterial pneumonia (VABP), or healthcare-associated bacterial pneumonia (HCABP)
* All subjects must fulfill at least 1 of the following clinical criteria at screening:

  1. New onset or worsening of pulmonary symptoms or signs, such as cough, dyspnea, tachypnea (eg, respiratory rate > 25 breaths/minute), expectorated sputum production, or requirement for mechanical ventilation
  2. Hypoxemia (eg, a partial pressure of oxygen [PaO2] < 60 mm Hg while the subject is breathing room air, as determined by arterial blood gas [ABG], or worsening of the ratio of the PaO2 to the fraction of inspired oxygen [PaO2/FiO2])
  3. Need for acute changes in the ventilator support system to enhance oxygenation, as determined by worsening oxygenation (ABG or PaO2/FiO2) or needed changes in the amount of positive end-expiratory pressure
  4. New onset of or increase in (quantity or characteristics) suctioned respiratory secretions, demonstrating evidence of inflammation and absence of contamination
* All subjects must have at least 1 of the following signs:

  1. Documented fever (ie, core body temperature [tympanic, rectal, esophageal] ≥ 38°C [100.4°F], oral temperature ≥ 37.5°C, or axillary temperature ≥ 37°C)
  2. Hypothermia (ie, core body temperature [tympanic, rectal, esophageal] ≤ 35°C [95.0°F], oral temperature ≤ 35.5°C and axillary temperature ≤ 36°C)
  3. Leukocytosis with a total peripheral white blood cell (WBC) count ≥ 10,000 cells/mm³
  4. Leukopenia with total peripheral WBC count ≤ 4500 cells/mm³
  5. Greater than 15% immature neutrophils (bands) noted on peripheral blood smear
* All subjects must have a chest radiograph during screening showing the presence of new or progressive infiltrate(s) suggestive of bacterial pneumonia. A computed tomography (CT) scan in the same time window showing the same findings could also be acceptable
* All subjects must have a suspected Gram-negative infection involving the lower respiratory tract

Exclusion Criteria:

* Subjects who have known or suspected community-acquired bacterial pneumonia (CABP), atypical pneumonia, viral pneumonia, or chemical pneumonia (including aspiration of gastric contents, inhalation injury)
* Other exclusions based on the prescribing information of meropenem or linezolid, prior antibiotic usage, age, and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (102):
- United States (15):
  - Shionogi Research Site, New Haven, Connecticut
  - Shionogi Research Site, DeLand, Florida
  - Shionogi Research Site, Chicago, Illinois
  - Shionogi Research Site, Council Bluffs, Iowa
  - Shionogi Research Site, Louisville, Kentucky
  - Shionogi Research Site, Baton Rouge, Louisiana
  - Shionogi Research Site, Shreveport, Louisiana
  - Shionogi Research Site, Annapolis, Maryland
  - Shionogi Research Site, Detroit, Michigan
  - Shionogi Research Site, St Louis, Missouri
  - Shionogi Research Site, Cleveland, Ohio
  - Shionogi Research Site, Columbus, Ohio
  - Shionogi Research Site, Bethlehem, Pennsylvania
  - Shionogi Research Site, Philadelphia, Pennsylvania
  - Shionogi Research Site, Salt Lake City, Utah
- Shionogi Research Site, Brussels, Belgium
- Canada (2):
  - Shionogi Research Site, Halifax, Nova Scotia
  - Shionogi Research Site, Kingston, Ontario
- Czechia (7):
  - Shionogi Research Site, Brno
  - Shionogi Research Site, Hradec Králové
  - Shionogi Research Site, Kolín
  - Shionogi Research Site, Kyjov
  - Shionogi Research Site, Ostrava-Poruba
  - Shionogi Research Site, Prague
  - Shionogi Research Site, Příbram
- Estonia (4):
  - Shionogi Research Site, Kohtla-Järve
  - Shionogi Research Site, Pärnu
  - Shionogi Research Site, Tallinn
  - Shionogi Research Site, Tartu
- France (7):
  - Shionogi Research Site, Angers
  - Shionogi Research Site, Argenteuil
  - Shionogi Research Site, Bron
  - Shionogi Research Site, LaRoche-sur-Yon
  - Shionogi Research Site, Lyon
  - Shionogi Research Site, Nice
  - Shionogi Research Site, Paris
- Georgia (3):
  - Shionogi Research Site, Batumi
  - Shionogi Research Site, Kutaisi
  - Shionogi Research Site, Tbilisi
- Germany (4):
  - Shionogi Research Site, Bonn
  - Shionogi Research Site, Hamburg
  - Shionogi Research Site, Heidelberg
  - Shionogi Research Site, Leipzig
- Hungary (4):
  - Shionogi Research Site, Budapest
  - Shionogi Research Site, Debrecen
  - Shionogi Research Site, Fehérgyarmat
  - Shionogi Research Site, Székesfehérvár
- Israel (5):
  - Shionogi Research Site, Holon
  - Shionogi Research Site, Jerusalem
  - Shionogi Research Site, Tel Aviv
  - Shionogi Research Site, Tel Litwinsky
  - Shionogi Research Site, Tikva
- Japan (6):
  - Shionogi Research Site, Maebashi, Gunma
  - Shionogi Research Site, Tsuchiura, Ibaraki
  - Shionogi Research Site, Tsu, Mie-ken
  - Shionogi Research Site, Shimajiri-gun, Okinawa
  - Shionogi Research Site, Itabashi-ku, Tokyo
  - Shionogi Research Site, Kumamoto
- Latvia (4):
  - Shionogi Research Site, Daugavpils
  - Shionogi Research Site, Liepāja
  - Shionogi Research Site, Riga
  - Shionogi Research Site, Saldus Novads
- Philippines (7):
  - Shionogi Research Site, Jaro, Iloilo City
  - Shionogi Research Site, Tondo, Manila
  - Shionogi Research Site, Caloocan, National Capital Region
  - Shionogi Research Site, Quezon City, National Capital Region
  - Shionogi Research Site, Caloocan
  - Shionogi Research Site, Iloilo City
  - Shionogi Research Site, Manila
- Shionogi Research Site, San Juan, Puerto Rico
- Russia (9):
  - Shionogi Research Site, Barnaul
  - Shionogi Research Site, Chelyabinsk
  - Shionogi Research Site, Krasnodar
  - Shionogi Research Site, Moscow
  - Shionogi Research Site, Novosibirsk
  - Shionogi Research Site, Saint Petersburg
  - Shionogi Research Site, Sait-Petersburg
  - Shionogi Research Site, Smolensk
  - Shionogi Research Site, Tomsk
- Serbia (3):
  - Shionogi Research Site, Belgrade
  - Shionogi Research Site, Kamenitz
  - Shionogi Research Site, Kragujevac
- Spain (6):
  - Shionogi Research Site, Alicante
  - Shionogi Research Site, Barcelona
  - Shionogi Research Site, Madrid
  - Shionogi Research Site, Torrejón de Ardoz
  - Shionogi Research Site, Torrevieja
  - Shionogi Research Site, Valencia
- Taiwan (3):
  - Shionogi Research Site, New Taipei City
  - Shionogi Research Site, Taichung
  - Shionogi Research Site, Taipei
- Ukraine (11):
  - Shionogi Research Site, Chernivtsi
  - Shionogi Research Site, Dnipropetrovsk
  - Shionogi Research Site, Ivano-Frankivsk
  - Shionogi Research Site, Kharkiv
  - Shionogi Research Site, Kherson
  - Shionogi Research Site, Kiev
  - Shionogi Research Site, Kremenchuk
  - Shionogi Research Site, Poltava
  - Shionogi Research Site, Sumy
  - Shionogi Research Site, Vinnitsya
  - Shionogi Research Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nordmann P, Shields RK, Doi Y, Takemura M, Echols R, Matsunaga Y, Yamano Y. Mechanisms of Reduced Susceptibility to Cefiderocol Among Isolates from the CREDIBLE-CR and APEKS-NP Clinical Trials. Microb Drug Resist. 2022 Apr;28(4):398-407. doi: 10.1089/mdr.2021.0180. Epub 2022 Jan 24. PMID 35076335
- [Derived] Skaar EP, Echols R, Matsunaga Y, Menon A, Portsmouth S. Iron serum levels and iron homeostasis parameters in patients with nosocomial pneumonia treated with cefiderocol: post hoc analysis of the APEKS-NP study. Eur J Clin Microbiol Infect Dis. 2022 Mar;41(3):467-476. doi: 10.1007/s10096-021-04399-9. Epub 2022 Jan 13. PMID 35025025
- [Derived] Wenzler E, Butler D, Tan X, Katsube T, Wajima T. Pharmacokinetics, Pharmacodynamics, and Dose Optimization of Cefiderocol during Continuous Renal Replacement Therapy. Clin Pharmacokinet. 2022 Apr;61(4):539-552. doi: 10.1007/s40262-021-01086-y. Epub 2021 Nov 18. PMID 34792787
- [Derived] Wunderink RG, Matsunaga Y, Ariyasu M, Clevenbergh P, Echols R, Kaye KS, Kollef M, Menon A, Pogue JM, Shorr AF, Timsit JF, Zeitlinger M, Nagata TD. Cefiderocol versus high-dose, extended-infusion meropenem for the treatment of Gram-negative nosocomial pneumonia (APEKS-NP): a randomised, double-blind, phase 3, non-inferiority trial. Lancet Infect Dis. 2021 Feb;21(2):213-225. doi: 10.1016/S1473-3099(20)30731-3. Epub 2020 Oct 12. PMID 33058798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included participants with hospital-acquired bacterial pneumonia (HABP), ventilator-associated bacterial pneumonia (VABP), or healthcare-associated bacterial pneumonia (HCABP) caused by Gram-negative bacteria.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to either cefiderocol or meropenem. Randomization was performed by the stratified randomization method using infection diagnosis (HABP, VABP, and HCABP) and Acute Physiology and Chronic Health Evaluation II (APACHE II) score (≤ 15 and ≥ 16) as allocation factors.
Groups:
- Cefiderocol: Participants received 2 g cefiderocol administered intravenously every 8 hours for 7 to 14 days and 600 mg linezolid administered intravenously every 12 hours for at least 5 days.
- Meropenem: Participants received 2 g meropenem administered intravenously every 8 hours for 7 to 14 days and 600 mg linezolid administered intravenously every 12 hours for at least 5 days.
Period: Overall Study
Arm/Group | Cefiderocol | Meropenem
Started | 148 | 152
Received Treatment | 148 | 150
Completed | 106 | 112
Not Completed | 42 | 40
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Recovery | 0 | 1
Not completed — Death | 39 | 34
Not completed — Other - Miscellaneous | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefiderocol | Meropenem | Total
Number analyzed (Participants) | 148 | 150 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (14.5) | 65.6 (15.1) | 65.2 (14.8)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 65 | 58 | 123
  >= 65 years | 83 | 92 | 175
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 93
  Male | 101 | 104 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 140 | 139 | 279
  Unknown or Not Reported | 4 | 8 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 102 | 100 | 202
  Black or African American | 0 | 1 | 1
  Asian | 44 | 44 | 88
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 2 | 4 | 6
  Missing | 0 | 1 | 1
Region [Count of Participants; unit: Participants]
  North America | 6 | 6 | 12
  South America | 0 | 0 | 0
  Europe | 99 | 100 | 199
  Asia-Pacific | 43 | 44 | 87
Clinical Diagnosis [Count of Participants; unit: Participants] — HABP = hospital acquired bacterial pneumonia; HCABP = healthcare-associated bacterial pneumonia; VABP = ventilator-associated bacterial pneumonia
  Participants
    VABP | 60 | 65 | 125
    HABP | 60 | 61 | 121
    HCABP | 28 | 24 | 52
Acute Physiology and Chronic Health Evaluation II (APACHE II) Score [Count of Participants; unit: Participants] — Acute Physiology And Chronic Health Evaluation II is a severity-of-disease classification applied within 24 hours of admission of a patient to an intensive care unit (ICU). The APACHE II score consists of three parts: 12 acute physiological variables, age, and chronic health status. The range of the score is 0 to 71, where higher scores correspond to more severe disease and a higher risk of death.
  Participants
    <= 15 | 75 | 78 | 153
    16 - 19 | 32 | 26 | 58
    >= 20 | 41 | 46 | 87

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality Rate at Day 14
Description: The all-cause mortality (ACM) rate at Day 14 was calculated as the percentage of participants in each treatment group who experienced mortality, regardless of the cause, from the first infusion of study drug up to Day 14.
  The Modified Intent-to-Treat Population included all randomized participants who met either of the following criteria:
  * Evidence of Gram-negative infection of the lower respiratory tract based on a culture, Gram-stain, or other diagnostic test
  * Evidence of a lower respiratory tract infection but culture or other diagnostic tests did not provide a microbiologic diagnosis
Time Frame: From first dose of study drug to Day 14
Population: Modified Intent-to-Treat Population; participants with known survival status.
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 145 | 146
percentage of participants | 12.4 | 11.6
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Non-Inferiority — The study hypothesis was that the all-cause mortality rate at Day 14 in participants who received cefiderocol would be non-inferior to that in participants who received high-dose meropenem. The margin of non-inferiority was 12.5%. Non-inferiority was concluded if the upper bound of the 2-sided 95% confidence interval for the difference in mortality at Day 14 between the 2 treatment groups (cefiderocol - meropenem) was smaller than 12.5%; p = 0.0020, Cochran-Mantel-Haenszel; Treatment Difference = 0.8, 95% CI 2-sided [-6.6 to 8.2] — Treatment difference (cefiderocol - meropenem) was the adjusted estimate of the difference in the ACM rate at Day 14 based on Cochran-Mantel Haenszel weights using APACHE II score (≤ 15 and ≥ 16) as the stratification factor

2. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at Test of Cure (TOC)
Description: Lower respiratory tract specimens (eg, sputum, endotracheal aspiration [ETA], endobronchial culture specimens collected by bronchoalveolar lavage [BAL], or protected specimen brush [PSB], lung biopsy tissue, pleural effusions, etc) were sent to the local microbiology laboratory for isolation and identification of pathogens.
  Microbiological outcome by Baseline pathogen at TOC was determined by the sponsor as either Eradication, Persistence, or Indeterminate. Overall per-participant microbiological outcome was determined based on the individual microbiological outcomes for each Baseline pathogen.
  Eradication: Absence of all Baseline Gram-negative pathogens from an appropriate clinical specimen (sputum, tracheal aspirate, bronchoalveolar lavage (BAL) fluid, protected specimen brush, pleural fluid, or lung biopsy). If it was not possible to obtain an appropriate clinical culture, and the participant had a successful clinical outcome, the response was presumed as eradication.
Time Frame: Test of cure (7 days after end of treatment; equivalent to Study Day 14 to 21)
Population: Modified Intent-to-Treat Population; participants with non-missing Baseline pathogen data
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 124 | 127
percentage of participants | 47.6 | 48.0
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Superiority; Treatment Difference = -1.4, 95% CI 2-sided [-13.5 to 10.7] — Treatment difference (cefiderocol - meropenem) was the adjusted estimate of the difference in the eradication rate calculated using Cochran-Mantel-Haenszel weights based on infection diagnosis (HABP/VABP/HCABP), and APACHE II score (≤ 15 and ≥ 16)

3. Secondary Outcome: Percentage of Participants With Clinical Cure at Test of Cure
Description: Clinical outcome was assessed by the investigator as either Clinical Cure, Clinical Failure, or Indeterminate.
  Clinical Cure: Resolution or substantial improvement of Baseline signs and symptoms of pneumonia, including a reduction in Sequential Organ Failure Assessment (SOFA) and Clinical Pulmonary Infection Score (CPIS) scores, and improvement or lack of progression of chest radiographic abnormalities such that no additional antibacterial therapy was required for the treatment of the current infection.
Time Frame: Test of cure (7 days after the end of treatment; equivalent to Study Day 14 to 21)
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 145 | 147
percentage of participants | 64.8 | 66.7
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Superiority; Treatment Difference = -2.0, 95% CI 2-sided [-12.5 to 8.5] — Treatment difference (cefiderocol - meropenem) was the adjusted estimate of the difference in the cure rate calculated using Cochran-Mantel-Haenszel weights based on infection diagnosis (HABP/VABP/HCABP), and APACHE II score (≤ 15 and ≥ 16)

4. Secondary Outcome: Percentage of Participants With Clinical Cure at Early Assessment (EA)
Description: as for outcome 3
Time Frame: Early assessment (Day 3-4 after the start of treatment)
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 145 | 147
percentage of participants | 82.8 | 83.0
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Other; Treatment Difference = -0.3, 95% CI 2-sided [-8.8 to 8.2] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Participants With Clinical Cure at End of Treatment (EOT)
Description: as for outcome 3
Time Frame: End of treatment (Day 7 to 14)
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 145 | 147
percentage of participants | 77.2 | 81.0
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Other; Treatment Difference = -3.8, 95% CI 2-sided [-12.8 to 5.1] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Percentage of Participants With Sustained Clinical Cure at Follow-up (FU)
Description: Clinical outcome was assessed by the investigator at follow-up as either Sustained Clinical Cure, Relapse, or Indeterminate.
  Sustained Clinical Cure: Continued resolution or substantial improvement of Baseline signs and symptoms of pneumonia, such that no antibacterial therapy was required for the treatment of pneumonia in a participant assessed as cured at TOC.
Time Frame: Follow-up (14 days after the end of treatment; Day 21 to 28)
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 145 | 147
percentage of participants | 57.9 | 57.8
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Other; Treatment Difference = -0.1, 95% CI 2-sided [-10.9 to 10.8] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at Early Assessment
Description: Microbiological outcome by Baseline pathogen at Early Assessment was determined by the sponsor as either Eradication, Persistence, or Indeterminate. Overall per-participant microbiological outcome was determined based on the individual microbiological outcomes for each Baseline pathogen.
  Eradication: Absence of all Baseline Gram-negative pathogens from an appropriate clinical specimen (sputum, tracheal aspirate, BAL fluid, protected specimen brush, pleural fluid, or lung biopsy). If it was not possible to obtain an appropriate clinical culture, and the participant had a successful clinical outcome, the response was presumed as eradication.
Time Frame: Early Assessment, Days 3 to 4
Population: Modified Intent-to-Treat Population; participants with non-missing Baseline pathogens
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 124 | 127
percentage of participants | 41.9 | 53.5
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Other; Treatment Difference = -12.4, 95% CI 2-sided [-24.4 to -0.5] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at End of Treatment
Description: Microbiological outcome by Baseline pathogen at End of Treatment was determined by the sponsor as either: Eradication, Persistence, or Indeterminate. Overall per-participant microbiological outcome was determined based on the individual microbiological outcomes for each Baseline pathogen.
  Eradication: Absence of all Baseline Gram-negative pathogens from an appropriate clinical specimen (sputum, tracheal aspirate, BAL fluid, protected specimen brush, pleural fluid, or lung biopsy). If it was not possible to obtain an appropriate clinical culture, and the participant had a successful clinical outcome, the response was presumed as eradication.
Time Frame: End of treatment, Day 7 to 14
Population: Modified Intent to-Treat Population; participants with non-missing Baseline pathogens
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 124 | 127
percentage of participants | 63.7 | 66.9
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Other; Treatment Difference = -3.8, 95% CI 2-sided [-15.5 to 7.9] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Percentage of Participants With Sustained Microbiologic Eradication at Follow-up
Description: Microbiological outcome by Baseline pathogen at Follow-up was determined by the sponsor as either Sustained Eradication, Persistence, Recurrence, or Indeterminate. Overall per-participant microbiological outcome was determined based on the individual microbiological outcomes for each Baseline pathogen.
  Sustained eradication: Absence of all Baseline Gram-negative pathogens from an appropriate clinical specimen (sputum, tracheal aspirate, BAL fluid, protected specimen brush, pleural fluid, or lung biopsy) after TOC. If it was not possible to obtain an appropriate clinical culture and the participant had a successful clinical response after TOC, the response was presumed to be eradication.
Time Frame: Follow-up (14 days after the end of treatment, Days 21 to 28)
Population: Modified Intent-to-Treat Population; participants with non-missing Baseline pathogens
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 124 | 127
percentage of participants | 43.5 | 38.6
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Other; Treatment Difference = 3.9, 95% CI 2-sided [-7.9 to 15.8] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: All-cause Mortality Rate at Day 28
Description: The all-cause mortality (ACM) rate at Day 28 was calculated as the percentage of participants who experienced mortality, regardless of the cause, from the first dose of study drug up to Day 28.
Time Frame: From first dose of study drug to Day 28
Population: Modified Intent-to-Treat Population; participants with known survival status.
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 143 | 146
percentage of participants | 21.0 | 20.5
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Other; Treatment Difference = 0.5, 95% CI 2-sided [-8.7 to 9.8] — Treatment difference (cefiderocol - meropenem) was the adjusted estimate of the difference in the ACM rate at Day 28 based on Cochran-Mantel Haenszel weights using APACHE II score (≤ 15 and ≥ 16) as the stratification factor

11. Secondary Outcome: All-cause Mortality Rate at the End of Study
Description: The all-cause mortality rate during both the treatment and follow-up period (up to the end of study [EOS] visit) was calculated as the percentage of participants who experienced mortality, regardless of the cause, from the first infusion of study drug up to EOS. If a participant discontinued from the study before EOS and survival information was not available, then the survival status for this endpoint for the participant was considered unknown.
Time Frame: From first dose of study drug through end of study (28 days after end of treatment, up to 42 days)
Population: Modified Intent-to-Treat Population; participants with known survival status.
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 142 | 146
percentage of participants | 26.8 | 23.3
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Test type: Other; Treatment Difference = 3.6, 95% CI 2-sided [-6.3 to 13.4] — Treatment difference (cefiderocol - meropenem) was the adjusted estimate of the difference in the ACM rate at EOS based on Cochran-Mantel Haenszel weights using APACHE II score (≤ 15 and ≥ 16) as the stratification factor

12. Secondary Outcome: Total Hospitalization Time
Description: The length of hospital stay attributable to the study-qualifying infection.
Time Frame: From first dose of study drug to test of cure (7 days after end of treatment; equivalent to Study Day 14 to 21) and to follow-up (14 days after the end of treatment; Day 21 to 28)
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 145 | 147
days
  Test of Cure | 11.54 (7.81) | 11.47 (7.32)
  Follow-up | 13.49 (10.06) | 12.98 (9.59)
Statistical Analysis 1: Comparison: Cefiderocol vs Meropenem; Comparison of Hospitalization time at test of cure; Test type: Superiority; p = 0.9382, t-test, 2 sided
Statistical Analysis 2: Comparison: Cefiderocol vs Meropenem; Comparison of hospitalization time at follow-up; Test type: Superiority; p = 0.6552, t-test, 2 sided

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: The severity of each adverse event (AE) was graded by the investigator according to the following definitions:
  * Mild: A finding or symptom is minor and does not interfere with usual daily activities.
  * Moderate: The event causes discomfort and interferes with usual daily activity or affects clinical status.
  * Severe: The event causes an interruption of the participant's usual daily activities or has a clinically significant effect.
  The relationship of each AE to the study treatment was determined by the investigator based on whether the AE could be reasonably explained as having been caused by the study drug (treatment related AE [TRAE]).
  An SAE is defined as any AE occurring at any dose that resulted in any of the following outcomes:
  * Death
  * Life-threatening condition
  * Hospitalization or prolongation of existing hospitalization for treatment
  * Persistent or significant disability/incapacity
  * Congenital anomaly/birth defect
  * Other medically important condition
Time Frame: From first dose of study drug through the end of study, up to 42 days.
Population: The safety population included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cefiderocol | Meropenem
Number analyzed (Participants) | 148 | 150
Participants
  Any adverse event | 130 | 129
  Mild adverse events | 33 | 37
  Moderate adverse events | 41 | 47
  Severe adverse events | 56 | 45
  Treatment-related adverse events | 14 | 17
  Serious adverse events | 54 | 45
  Treatment-related serious adverse events | 3 | 5
  AEs leading to discontinuation of study drug | 12 | 14
  TRAE leading to discontinuation of study drug | 2 | 2
  Adverse events leading to death | 39 | 35

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of study, up to 42 days.
Arm/Group | Cefiderocol | Meropenem
All-Cause Mortality (participants affected / at risk) | 39/148 | 35/150
Serious Adverse Events (participants affected / at risk) | 54/148 | 45/150
Other Adverse Events (participants affected / at risk) | 119/148 | 123/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cefiderocol (N=148) | Meropenem (N=150)
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 7 | 5
Cardiac failure (Cardiac disorders) | 2 | 3
Cardiac failure acute (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 3 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 4 | 4
Sudden death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Meningoencephalitis bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 3
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 2
Septic encephalopathy (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 4 | 1
Spinal cord infection (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 5
Liver function test abnormal (Investigations) | 0 | 1
Liver function test increased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 5
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 2 | 1
Lacunar stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Stroke in evolution (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Leg amputation (Surgical and medical procedures) | 1 | 0
Femoral artery embolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cefiderocol (N=148) | Meropenem (N=150)
Anaemia (Blood and lymphatic system disorders) | 12 | 12
Thrombocytosis (Blood and lymphatic system disorders) | 4 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 6
Atrial fibrillation (Cardiac disorders) | 7 | 4
Bradycardia (Cardiac disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 13 | 13
Constipation (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 1 | 4
Pyrexia (General disorders) | 5 | 5
Oedema peripheral (General disorders) | 2 | 3
Hepatocellular injury (Hepatobiliary disorders) | 0 | 3
Urinary tract infection (Infections and infestations) | 22 | 15
Pneumonia (Infections and infestations) | 5 | 5
Clostridium difficile infection (Infections and infestations) | 4 | 3
Urinary tract infection fungal (Infections and infestations) | 4 | 2
Tracheobronchitis (Infections and infestations) | 2 | 4
Bronchitis (Infections and infestations) | 2 | 3
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 9 | 5
Alanine aminotransferase increased (Investigations) | 8 | 6
Gamma-glutamyltransferase increased (Investigations) | 5 | 2
Transaminases increased (Investigations) | 4 | 3
Hepatic enzyme increased (Investigations) | 3 | 5
Amylase increased (Investigations) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 16 | 23
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1
Gout (Metabolism and nutrition disorders) | 1 | 3
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 3
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 4
Headache (Nervous system disorders) | 3 | 1
Delirium (Psychiatric disorders) | 5 | 4
Insomnia (Psychiatric disorders) | 5 | 3
Anxiety (Psychiatric disorders) | 3 | 0
Agitation (Psychiatric disorders) | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 | 10
Hypertension (Vascular disorders) | 5 | 7
Phlebitis (Vascular disorders) | 3 | 4
Hypotension (Vascular disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT03032380/SAP_000.pdf
  • Study Protocol (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT03032380/Prot_001.pdf